CLINICAL TRIAL: NCT00219401
Title: Neonatal Immunization With Pneumococcal Conjugate Vaccine in Papua New Guinea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: The University of Western Australia (Other)
Responsible Party: A/Prof. Deborah Lehmann, University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 071613/Z/03/Z; 303123 NHMRC Australia
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Pneumonia; Meningitis; Otitis Media
Keywords: Pneumococcal vaccine; Antibody responses; Cellular immunology; Th1/Th2 immune responses; Paediatric; Neonatal; Infectious diseases; Papua New Guinea
MeSH Terms: conditions — Pneumonia; Meningitis; Otitis Media; Communicable Diseases | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neonatal 7vPCV (Experimental): Receive study vaccine (Prevnar) at birth, 1 and 2 months
  Interventions: Biological: Pneumococcal 7 valent conjugate vaccine (Prevenar®)
- Infant 7vPCV (Experimental): Receive the study vaccine (Prevnar) at 1, 2 and 3 months
  Interventions: Biological: Pneumococcal 7 valent conjugate vaccine (Prevenar®)
- Control (Placebo Comparator): Do not receive study vaccine (Prevnar)
  Interventions: Biological: Pneumococcal 7 valent conjugate vaccine (Prevenar®)

INTERVENTIONS:
Biological: Pneumococcal 7 valent conjugate vaccine (Prevenar®) — Accelerated PCV vaccinaton.

SUMMARY:
The National Health Plan 2001-2010 calls for investigation of the feasibility of pneumococcal vaccines for Papau New Guinea. The Papua New Guinea (PNG) Institute of Medical Research, the Telethon Institute for Child Health Research and the Department of Paediatrics, University of Western Australia will collaborate to examine very closely the safety of neonatal vaccination, particularly with regard to impact on the development of immunity and response to other vaccines given to infants. This study will also provide a unique opportunity for training of PNG and Australian scientists in both countries.

DETAILED DESCRIPTION:
In order to obtain the earliest possible protection against invasive pneumococcal disease, achieve optimal coverage and reduce burden of early carriage, neonatal pneumococcal conjugate vaccine (PCV) immunization needs to be considered. This study in the PNG highlands will enrol 312 infants at birth, who will be randomised to receive PCV either at 1-2-3 months (infant schedule according to PNG national EPI schedule) or 0-1-2 months of age (neonatal schedule) or receive only routine immunizations (controls). Blood samples will be taken at birth-2-3-4 months of age, pre- and post-pneumococcal polysaccharide booster (23vPPV) at 9-10 months of age (to assess immune memory) and at 18 months at study completion. Carriage will be assessed weekly for the first month of life and at regular intervals thereafter. There will be ongoing surveillance for respiratory and other diseases throughout the study. In addition to serotype-specific IgG, we will examine IgG avidity, IgG subclasses, mucosal IgA and T-cell cytokine responses to PCV and pneumococcal protein antigens. To ensure immunological safety, particularly for neonatal PCV, immune responses to concomitant vaccines and viral and environmental antigens will also be examined as well as overall T-cell maturation.

ELIGIBILITY:
Inclusion Criteria:

New born babies with birth weight >2000 g (2 kgs) and parents giving consent

Exclusion Criteria:

1. Acute neonatal infection;
2. Severe congenital abnormality;
3. Children of mothers known to be HIV positive will be excluded;
4. Serious asphyxia at birth;
5. Intended migration in the next 2 years;
6. Parents withdraw consent;

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity and Safety | 5 yrs
  Serum PCV serotype-specific IgG antibody at 2, 4 and 9 mths. Mucosal PCV serotype-specific IgG antibody at 1, 3, 4 and 9 mths. PCV-induced T-cell memory (against vaccine protein carrier) at 3 and 9 mths. Local and systemic reactogenicity 48-96 hrs after vaccination. Monitoring of serious adverse events during 18 mth follow-up. T-cell development to bystander antigens at 3 and 9 mths.

SECONDARY OUTCOMES:
Immunogenicity | 5 years
  Serum PCV and non-PCV serotype specific IgG antibody at 10 mths, after 23vPPV vaccination at 9 mths
Pneumococcal-specific acquired immunity | 5 years
  Assessment of cellular immune responses to pneumococcal protein antigens at 9 and 18 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siba, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research; Deborah Lehmann, MBBS, Msc, Principal Investigator — Telethon Institute for Child Health Research
Locations (1):
- Papua New Guinea Institute of Medical Research, Goroka, EHP, Papua New Guinea

REFERENCES:
- [Result] van den Biggelaar AH, Richmond PC, Pomat WS, Phuanukoonnon S, Nadal-Sims MA, Devitt CJ, Siba PM, Lehmann D, Holt PG. Neonatal pneumococcal conjugate vaccine immunization primes T cells for preferential Th2 cytokine expression: a randomized controlled trial in Papua New Guinea. Vaccine. 2009 Feb 25;27(9):1340-7. doi: 10.1016/j.vaccine.2008.12.046. Epub 2009 Jan 14. PMID 19150378
- [Result] van den Biggelaar AH, Pomat W, Bosco A, Phuanukoonnon S, Devitt CJ, Nadal-Sims MA, Siba PM, Richmond PC, Lehmann D, Holt PG. Pneumococcal conjugate vaccination at birth in a high-risk setting: no evidence for neonatal T-cell tolerance. Vaccine. 2011 Jul 26;29(33):5414-20. doi: 10.1016/j.vaccine.2011.05.065. Epub 2011 Jun 7. PMID 21645573
- [Result] Francis JP, Richmond PC, Pomat WS, Michael A, Keno H, Phuanukoonnon S, Nelson JB, Whinnen M, Heinrich T, Smith WA, Prescott SL, Holt PG, Siba PM, Lehmann D, van den Biggelaar AH. Maternal antibodies to pneumolysin but not to pneumococcal surface protein A delay early pneumococcal carriage in high-risk Papua New Guinean infants. Clin Vaccine Immunol. 2009 Nov;16(11):1633-8. doi: 10.1128/CVI.00247-09. Epub 2009 Sep 23. PMID 19776196
- [Derived] van den Biggelaar AHJ, Richmond PC, Fuery A, Anderson D, Opa C, Saleu G, Lai M, Francis JP, Alpers MP, Pomat WS, Lehmann D. Pneumococcal responses are similar in Papua New Guinean children aged 3-5 years vaccinated in infancy with pneumococcal polysaccharide vaccine with or without prior pneumococcal conjugate vaccine, or without pneumococcal vaccination. PLoS One. 2017 Oct 13;12(10):e0185877. doi: 10.1371/journal.pone.0185877. eCollection 2017. PMID 29028802
- [Derived] Francis JP, Richmond PC, Michael A, Siba PM, Jacoby P, Hales BJ, Thomas WR, Lehmann D, Pomat WS, van den Biggelaar AHJ. A longitudinal study of natural antibody development to pneumococcal surface protein A families 1 and 2 in Papua New Guinean Highland children: a cohort study. Pneumonia (Nathan). 2016 Aug 15;8:12. doi: 10.1186/s41479-016-0014-x. eCollection 2016. PMID 28702291
- [Derived] Aho C, Michael A, Yoannes M, Greenhill A, Jacoby P, Reeder J, Pomat W, Saleu G, Namuigi P, Phuanukoonnon S, Smith-Vaughan H, Leach AJ, Richmond P, Lehmann D; Neonatal Pneumococcal Conjugate Vaccine Trial Study Team. Limited impact of neonatal or early infant schedules of 7-valent pneumococcal conjugate vaccination on nasopharyngeal carriage of Streptococcus pneumoniae in Papua New Guinean children: A randomized controlled trial. Vaccine Rep. 2016 Dec;6:36-43. doi: 10.1016/j.vacrep.2016.08.002. PMID 28580433
- [Derived] Pomat WS, van den Biggelaar AH, Phuanukoonnon S, Francis J, Jacoby P, Siba PM, Alpers MP, Reeder JC, Holt PG, Richmond PC, Lehmann D; Neonatal Pneumococcal Conjugate Vaccine Trial Study Team. Safety and immunogenicity of neonatal pneumococcal conjugate vaccination in Papua New Guinean children: a randomised controlled trial. PLoS One. 2013;8(2):e56698. doi: 10.1371/journal.pone.0056698. Epub 2013 Feb 22. PMID 23451070